CLINICAL TRIAL: NCT02785926
Title: Impact of Antenatal Exposure to Pesticides on Neurophysiological Functions (Sleep, Respiration) of Preterm Neonates
Acronym: PHYSIOMECO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0018
Record Dates: First submitted 2016-05-23; First posted 2016-05-30 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Premature Infants
Keywords: pesticide exposure; respiratory control; sleep
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
During pregnancy, the foetus is therefore chronically exposed to a large number of substances. A number of studies have started to emphasize the effects of this antenatal exposure on the newborn infant's morphological parameters (weight, crown-rump length, etc.). However, in addition to these morphological effects, pesticides may also induce various effects on physiological functions, as some pesticides act as inhibitors of neurotransmitters involved in many nervous system regulation pathways in man. This is particularly the case for organophosphates, which act as acetylcholinesterase inhibitors. A previous study conducted by the coordinator of the project presented here demonstrated the presence of high levels of this type of pesticide in meconium (1st stool) in neonates born in Picardy. This inhibition of the enzyme metabolizing ACh could have an impact on neurophysiological functions mediated by this neurotransmitter. Sleep or respiratory control, vital functions of the neonate particularly in preterm neonates, could therefore be affected.

The PhysioMéco project is therefore designed to study the possible links between antenatal exposure to pesticides and modifications of respiratory control allowed by peripheral chemoreceptor in preterm neonates. Antenatal exposure will be determined by pesticide assays in the meconium of neonates in combination with an exposure questionnaire to determine the sources of these pesticides. Sleep and respiratory control will be studied in these neonates nursed in incubators. Hypoxic test will be used in order to assess respiratory control involving the peripheral chemoreceptors.

ELIGIBILITY:
Inclusion Criteria:

* premature neonates born at after 26 week of gestational age studied after 32 weeks, mothers living in Picardy and more than 18 years

Exclusion Criteria:

* neonates with neurological, respiratory and cardiac disorders or receiving treatments known to affect cardiorespiratory variables or sleep structure

Ages: 26 Weeks to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature neonates
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
response to hypoxia test (i.e peripheral chemoreceptor activity) in exposed and no exposed premature infant | 10 days

SECONDARY OUTCOMES:
arousal in response to hypoxic test | 10 weeks
sleep structure with EEG | 10 weeks
apnea frequency | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: André LEKE, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France